CLINICAL TRIAL: NCT04367727
Title: Effect of Different Pre Application Time Intervals of Light Emitting Diode Therapy on Muscle
Brief Title: Effect of Light Emitting Diode Therapy on Muscle Fatigue
Acronym: LED
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, HAhmed, Principal investigator, Cairo University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: P.T.REC/012/002480
Record Dates: First submitted 2020-01-24; First posted 2020-04-29 (Actual); Last update posted 2020-11-25 (Actual); Status verified 2020-11

CONDITIONS: Muscle Fatigue

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- 5 minutes before 1 (Experimental): Light emitting diode applied 5 minutes before fatiguing task
  Interventions: Device: Light emitting diode
- 5 minutes before 2 (Placebo Comparator): Light emitting diode applied 5 minutes before fatiguing task
  Interventions: Device: Light emitting diode
- 1 hour before 1 (Experimental): Light emitting diode applied 1 hour before fatiguing task
  Interventions: Device: Light emitting diode
- 1 hour before 2 (Placebo Comparator): Light emitting diode applied 1 hour before fatiguing task
  Interventions: Device: Light emitting diode
- 5 hours before 1 (Experimental): Light emitting diode applied 5 hours before fatiguing task
  Interventions: Device: Light emitting diode
- 5 hours before 2 (Placebo Comparator): Light emitting diode applied 5 hours before fatiguing task
  Interventions: Device: Light emitting diode

INTERVENTIONS:
Device: Light emitting diode — Light emitting diode at a wavelength of 890 nm is produced by an array of 60 gallium aluminum arsenide light-emitting diodes located on flexible pads and the near infrared photo energy is delivered in a noninvasive, drug-free manner

SUMMARY:
The purpose of this study is to determine the optimal time interval between light emitting diode application and exercise to improve fatigue resistance.The results of this study could be useful in planning a rehabilitation program in musculature disorders and also in athletic training.

DETAILED DESCRIPTION:
1. To determine the effect of light emitting diode applied 5 minutes before exercise on pain, rate of perceived exertion and maximum voluntary contraction.
2. To determine the effect of light emitting diode applied 1 hour before exercise on pain, rate of perceived exertion and maximum voluntary contraction.
3. To determine the effect of light emitting diode applied 5 hours before exercise on pain, rate of perceived exertion and maximum voluntary contraction.
4. To determine the difference between light emitting diode applied 5 minutes,1 hour or 5 hours before exercise on pain, rate of perceived exertion and maximum voluntary contraction.

ELIGIBILITY:
Inclusion Criteria:

* Healthy non athletics subjects.
* Age ranges from 20-40 years.
* Body mass index is less than 25 kg/m 2

Exclusion Criteria:

* Neurological deficit and recent injury to either upper extremity
* non diagnosed pain .
* Contraindications to LED irradiation (such as light hypersensitivity, fluctuating blood pressure, insufficient blood circulation, fever and inflammation of the skin)
* Conditions in which physical exertion is contraindicated (such as cardiovascular deficits, hypertension and respiratory problems)
* Restriction in shoulder or elbow range of motion;
* Neoplasm,
* Rheumatoid,
* Strength training in the past 6 months;
* Previous surgery in the spine or upper extremity;
* Complaints of pain in the shoulder, elbow,wrist, and trunk musculature system;
* Use of dietary supplements; and not in any other exercise program for at least the past 3 months.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-01 (Estimated); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
Isometric peak torque of elbow flexors | change from before light emitting diode application at 5 minutes, 1 hour and 5 hours
  metric unit is Newton
Isometric peak torque of elbow flexors | change from before light emitting diode application at1 minute
  metric unit is Newton
Isokinetic peak torque of elbow flexors | change from before light emitting diode application at 5 minutes, 1 hour and 5 hours
  Metric unit is Newton and at angular velocity 60
Isokinetic peak torque of elbow flexors | change from before light emitting diode application at 1 minute after light emitting diode application
  Metric unit is Newton and at angular velocity 60

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Physical Therapy, Cairo, Egypt